CLINICAL TRIAL: NCT01503489
Title: Risk for Antidepressant-associated Switch From Depression to Hypomania, Mania, or Mixed Episode During the 8 Weeks After the Introduction of an Antidepressant or After Increasing the Dosage of Baseline Antidepressant.
Brief Title: Risk Factors for AD-Associated Switch to Mania
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Professor Eduard Vieta Pascual, MD, Psychiatrist, PhD, MD, PhD, Hospital Clinic of Barcelona
Other Study IDs: SWITCH.
Record Dates: First submitted 2011-12-29; First posted 2012-01-04 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Bipolar Disorder
Keywords: Switch
MeSH Terms: conditions — Bipolar Disorder | interventions — Selective Serotonin Reuptake Inhibitors; Antidepressive Agents, Tricyclic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bipolar depressed patients: Bipolar I or II outpatients, current major depressive episode (HDRS-17 over 20).
  Interventions: Drug: Selective Serotonin Reuptake Inhibitors (SSRI), Serotonin-Norepinephrine Reuptake Inhibitor( SNRI), and Tricyclics.

INTERVENTIONS:
Drug: Selective Serotonin Reuptake Inhibitors (SSRI), Serotonin-Norepinephrine Reuptake Inhibitor( SNRI), and Tricyclics. — Risk for antidepressant-associated switch from depression to hypomania, mania, or mixed episode during the 8 weeks after the introduction of an antidepressant or after increasing the dosage of baseline antidepressant.
  Other Names: Selective Serotonin Reuptake Inhibitors; Serotonin-Norepinephrine Reuptake Inhibitor; Tricyclics Antidepressants

SUMMARY:
The present study aimed at identifying clinical risk factors for switch into (hypo)mania or mixed states, within 8 weeks after introduction of an antidepressant or after increasing its dosage.

DETAILED DESCRIPTION:
Treatment of bipolar depression with antidepressants is strongly debated for the methodologically poor and insufficient data supporting their use and the widely held belief that antidepressants can induce new episodes of abnormal mood elevation or accelerate the rate of cycling. The present study aimed at identifying clinical risk factors for switch into (hypo)mania or mixed states, within 8 weeks after introduction of an antidepressant or after increasing its dosage, in a prospective, longitudinal design.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I and II disorder.

Exclusion Criteria:

* Major medical comorbidities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bipolar I and II disorder patients.
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Risk for antidepressant-associated switch from depression to hypomania, mania, or mixed episode during the 8 weeks after the introduction of an antidepressant or after increasing the dosage of baseline antidepressant. | 8 weeks.
  Bipolar I or II outpatients, current major depressive episode (HDRS-17 over 20), were treated with any antidepressant combined with treatment-as-usual, as decided by the treating psychiatrist.
  Treatment-emergent affective switch was defined as fully syndromic hypomanic, manic, or mixed episode: YMRS >12 and an increase of 5 points or more compared to the last assessment for hypomanic/manic features, and YMRS and HDRS-17 >14 for a mixed episode.
  The above-mentioned alterations needed to occur within 8 weeks after introduction of the antidepressant or after increasing the dosage.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Valenti, MD, Study Director — Bipolar Disorders Program, Hospital Clinic Barcelona.
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Valenti M, Pacchiarotti I, Undurraga J, Bonnin CM, Popovic D, Goikolea JM, Torrent C, Hidalgo-Mazzei D, Colom F, Vieta E. Risk factors for rapid cycling in bipolar disorder. Bipolar Disord. 2015 Aug;17(5):549-59. doi: 10.1111/bdi.12288. Epub 2015 Feb 12. PMID 25682854
- [Derived] Valenti M, Pacchiarotti I, Bonnin CM, Rosa AR, Popovic D, Nivoli AM, Goikolea JM, Murru A, Undurraga J, Colom F, Vieta E. Risk factors for antidepressant-related switch to mania. J Clin Psychiatry. 2012 Feb;73(2):e271-6. doi: 10.4088/JCP.11m07166. PMID 22401488